CLINICAL TRIAL: NCT03152370
Title: An Open-Label Multicenter Phase 1b Study of E7046 in Combination With Radiotherapy/Chemoradiotherapy (RT/CRT) in Preoperative Treatment of Subjects With Rectum Cancer
Brief Title: Preoperative Radiotherapy and E7046 in Rectum Cancer
Acronym: PRAER 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adlai Nortye Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7046-G000-102; 2016-003064-38 (EudraCT Number)
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Neoadjuvant Therapy in Rectal Cancer
Keywords: E7046; Radiotherapy/Chemoradiotherapy; Neoadjuvant therapy; Rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — E7046; Capecitabine

STUDY DESIGN:
Intervention Model Description: This study will investigate two neoadjuvant radiotherapy/chemoradiotherapy schedules in combination with E7046 in parallel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- E7046 in combination with Long Course Chemoradiotherapy (LCRT) (Experimental): Participants will receive once daily (QD) doses of E7046 (recommended Phase 2 dose [RP2D] determined in the Dose-Escalation part of the study) for 10 weeks, starting on Day 1, 14 days prior to initiation of the radiotherapy. LCRT will be initiated on Day 15 and will consist of a total of 45 Grays (GY) radiation administered in 1.8 GY daily doses delivered for 5 days (Monday to Friday) every week for 5 weeks. Capecitabine (825 milligrams per meters squared [mg/m^2]) will be administered twice daily on the days of radiotherapy. Surgery will be performed 14 to 16 weeks from the first day of E7046 treatment.
  Interventions: Drug: E7046; Radiation: Long Course Chemoradiotherapy (LCRT); Drug: capecitabine
- E7046 in combination with SCRT followed by chemotherapy (Experimental): Participants will receive QD doses of E7046 (RP2D determined in the Dose-Escalation part of the study) for 10 weeks, starting on Day 1, 14 days prior to initiation of the radiotherapy. Short course radiotherapy (SCRT) will be initiated on Day 15 and will consist of a total of 25 Gy radiation administered in 5 Gy daily doses for 5 days (Monday to Friday) for 1 week. Ten days after the end of radiotherapy, 3 cycles of the modified folinic acid/5-FU/oxaliplatin (mFOLFOX-6) regimen will be administered every 2 weeks for 2 consecutive days. Surgery will be performed 14 to 16 weeks from the first day of E7046 treatment.
  Interventions: Drug: E7046; Radiation: Short Course Radiotherapy (SCRT); Drug: folinic acid/5-FU/oxaliplatin (mFOLFOX-6)

INTERVENTIONS:
Drug: E7046 — oral administration
Radiation: Long Course Chemoradiotherapy (LCRT) — pelvic radiotherapy
  Arms: E7046 in combination with Long Course Chemoradiotherapy (LCRT)
Radiation: Short Course Radiotherapy (SCRT) — pelvic radiotherapy
  Arms: E7046 in combination with SCRT followed by chemotherapy
Drug: capecitabine — chemotherapy
  Arms: E7046 in combination with Long Course Chemoradiotherapy (LCRT)
Drug: folinic acid/5-FU/oxaliplatin (mFOLFOX-6) — chemotherapy
  Arms: E7046 in combination with SCRT followed by chemotherapy

SUMMARY:
This is a multicenter, open-label, Phase 1b study in participants with locally advanced rectum cancer where primary resection without chemoradiotherapy is unlikely to achieve clear margins as defined by magnetic resonance imaging (MRI). It is conducted to assess the safety, to assess the tolerability, and to determine the recommended Phase 2 dose (RP2D) of E7046 in combination with pre-operative chemoradiotherapy. The study will also assess the efficacy of the combination in the expansion part at RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed invasive primary rectal carcinoma
* Age ≥18 years at the time of informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Participants must have locally advanced rectum cancer where primary resection without chemoradiotherapy (CRT) is unlikely to achieve clear margins as defined by magnetic resonance imaging (MRI), with no metastatic disease, as assessed by independent review.
* Disease that can be encompassed within a radical radiotherapy treatment volume
* Participant must consent to repeated biopsy to allow the acquisition of fresh and/or formalin-fixed paraffin-embedded (FFPE) material. Available archived tumor material may be submitted as the pretreatment biopsy provided that minimum requirements are met by local pathology review as defined in the laboratory manual. If archived tumor material is not available or does not meet minimum requirements, then a fresh tumor biopsy must be obtained in accordance with local institutional practice.
* Adequate renal function defined as serum creatinine <1.5 × upper limit of normal (ULN) (or use System of Units [SI] units or calculated creatinine clearance ≥50 milliliter per minute [mL/min] per the Cockcroft and Gault formula)
* Adequate bone marrow function:

  * Absolute neutrophil count (ANC) ≥1500/millimeters cubed (mm^3) (≥1.5 × 10^3/microliters [µL])
  * Platelets ≥100,000/mm^3 (≥100 × 10^9/Liters [L])
  * Hemoglobin ≥9.0 grams per deciliter (g/dL)
* Adequate liver function:

  * Adequate blood coagulation function as evidenced by an International Normalized Ratio (INR) ≤1.5
  * Total bilirubin ≤1.5 × ULN except for unconjugated hyperbilirubinemia or Gilbert's syndrome
  * Alkaline phosphatase, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) ≤2.5 × ULN
* No prior pelvic radiotherapy, chemotherapy, immunotherapy, or other anti-cancer treatment for rectal cancer
* No prior exposure to colony stimulating factor 1 receptor (CSF1R) antagonists such as but not limited to emactuzumab (RG7155) (Roche), PLX3397 (Plexicon), JNJ40346627 (Johnson & Johnson), including both anti-CSF1R and small molecule inhibitors and prostaglandin E2 receptor 4 (EP4) antagonists
* No preexisting condition that would deter radiotherapy, eg, fistulas, severe ulcerative colitis (particularly participants currently taking sulphasalazine), Crohn's disease, prior adhesions
* Willing and able to give informed consent and comply with all aspects of the protocol

Exclusion Criteria:

* Any contraindications to MRI (eg, participants with pacemakers, claustrophobia, excessive weight, etc).
* Unfit to receive study treatment or subsequent surgical resection
* Active hydronephrosis
* Unequivocal evidence of metastatic disease defined by computerized tomography (CT) (includes resectable metastases)
* Prolongation of corrected QT (QTc) interval to >480 milliseconds (msec) when electrolyte balance is normal
* Recent occurrence (within 3 to 6 months) of a major thromboembolic event, such as pulmonary embolism or proximal deep vein thrombosis, unless stable on (>1 month) therapeutic anticoagulation (aspirin <325 milligrams (mg) daily or low-molecular-weight heparin [LMWH]). Participants with a history of clinically non-significant thromboembolic events, not requiring anticoagulation, are allowed on study.
* Participants receiving oral warfarin are not eligible for this study (unless warfarin is discontinued at least 7 days prior to commencement of treatment and for the duration of the study, or oral warfarin is converted to LMWH, where local clinical opinion considers this an acceptable option).
* Previous radiotherapy in the pelvic region (eg, prostate) or previous rectal surgery (eg, total mesorectal excision [TME]) or any investigational treatment for rectal cancer
* Cardiac conditions as follows: uncontrolled hypertension (resting blood pressure [BP] ≥150/95 millimeters of mercury [mmHg] despite optimal therapy), heart failure New York Heart Association (NYHA) Class II or above, prior or current cardiomyopathy, atrial fibrillation with heart rate >100 beats per minute (bpm). Unstable ischemic heart disease (myocardial infarction within 6 months prior to starting treatment, or angina requiring use of nitrates more than once weekly)
* Has a known additional malignancy that is progressing and/or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy, previous ductal carcinoma in situ (DCIS), or breast cancer diagnosed more than 5 years ago, as long as adequately treated or in situ, or early (up to stage 1B1) cervical cancer, or vulval intraepithelial neoplasia (VIN), or vulval cancer adequately treated without pelvic radiation therapy (RT)
* Refractory nausea and vomiting, chronic gastrointestinal diseases (eg, inflammatory bowel disease), or significant bowel resection that may impair adequate absorption and bioavailability of study drug. Major disturbance of bowel function (eg, gross fecal incontinence or requiring >6 mg loperamide each day).
* Participants with prior Hepatitis B or C infection with inadequate liver function
* Recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access and defunctioning stoma or any other surgical procedures not considered major by the investigator) that would prevent administration of study treatment
* Known dihydropyrimidine dehydrogenase (DPD) deficiency
* Participants with progressive neurological dysfunction that would confound the evaluation of neurological and other toxicities; any evidence of severe or uncontrolled systemic disease, active infection, active bleeding diatheses or renal transplant, including any participant with known active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection
* Participants with interstitial pneumonia or extensive and symptomatic fibrosis of the lungs
* Participants with any active autoimmune disease or a documented history of autoimmune disease, poorly controlled asthma or history of syndrome that required systemic steroids or immunosuppressive medications, except for participants with vitiligo or resolved childhood asthma/atopy. Participants with asthma who require intermittent use of bronchodilators (such as albuterol) will not be excluded from this study.
* Any other major illness that, in the investigator's judgment, will substantially increase the risk associated with the participant's participation in this study
* Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (eg, Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [β-hCG] test with a minimum sensitivity of 25 International Units per Liter [IU/L] or equivalent units of ß-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug. Females of childbearing potential (all females will be considered to be of childbearing potential unless they are postmenopausal [amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause] or have been sterilized surgically [ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing]) who:

  * Had unprotected sexual intercourse within 30 days before study entry and who do not agree to use a highly effective method of contraception (eg, true abstinence if it is their preferred and usual lifestyle [defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments], an intrauterine device, a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 6 months after study drug discontinuation;
  * Are not currently abstinent or do not agree to refrain from sexual activity during the study period and for 6 months after study drug discontinuation;
  * Are using hormonal contraceptives but are not on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and who do not agree to use the same contraceptive during the study or for 6 months after study drug discontinuation.
* Males who have not had a successful vasectomy (confirmed azoospermia) or they and their female partners do not meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception throughout the study period or for 6 months after study drug discontinuation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose (MTD) in combination with pre-operative chemoradiotherapy | 10 weeks
  The MTD is defined as one dose level below the dose level where ≥2 of 6 participants experience a dose-limiting toxicity (DLT; study drug-related toxicity) (ie, ≥33% of participants with a DLT at that dose level).
Number of participants with DLTs | 10 weeks
  DLTs are defined as study drug-related toxicities meeting specified grades per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) 4.03.
Number of participants with any serious adverse event (SAE) | 10 weeks
  An SAE is any untoward medical occurrence that at any dose: results in death; is life threatening (ie, the participant was at immediate risk of death from the adverse event as it occurred; this does not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug).
Number of participants with any non-serious adverse event (AE) | 10 weeks
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with the medicinal product.

SECONDARY OUTCOMES:
Pathological complete response (pCR) rate | 14 to 16 weeks from the first dose of E7046
  pCR is defined as the absence of any viable tumor cell on the resected specimen, irrespective of the proportions of necrosis and fibrosis.
Number of participants with a histopathologically confirmed circumferential margin negative (CRM-ve) resection | 14 to 16 weeks from the first dose of E7046
  The circumferential resection margin in rectal cancer has been defined as the non-peritonealized surface of a resection specimen created by dissection of the subperitoneal aspect at surgery.
Number of participants with the indicated histopathologically confirmed tumor regression grade | 14 to 16 weeks from the first dose of E7046
  The pathologic tumor regression grade is defined as the tumor regression grade on posttreatment histopathological examination of the resection specimen.
Number of participants with the indicated magnetic resonance imaging (MRI)-confirmed tumor regression grade | 11 to 13 weeks after the first dose of E7046
  MRI-confirmed tumor regression grade is defined as the tumor regression grade on MRI images obtained after chemoradiotherapy.
Number of participants with the indicated MRI-confirmed down staging in T stage | 11 to 13 weeks after the first dose of E7046
  Downstaging in T stage is defined as a reduction in T stage after chemoradiotherapy on MRI images.
Disease-free survival (DFS) | up to 2 years
  Disease-free survival is defined as the time from treatment start to the date of the first documented disease occurrence, or date of death, whichever occurs first.
Mean maximum observed concentration (Cmax) for E7046 and its metabolite ER-888188 in plasma | Day 1, Day 8, Week 3, Week 7
  Dose-Escalation: Day 1 and Day 8 at predose (0 hours [hr]); 0.5, 1, 2, 4, 6, 8, 10, and 24 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose (from participants on E7046 treatment). Expansion Cohort: Day 1 and Day 8 at predose; 0.5 to 4 hr and 8 to 12 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose
Mean time at which the highest drug concentration (Tmax) occurs for E7046 and its metabolite ER-888188 in plasma | Day 1, Day 8, Week 3, Week 7
  Dose-Escalation: Day 1 and Day 8 at predose (0 hr); 0.5, 1, 2, 4, 6, 8, 10, and 24 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose (from participants on E7046 treatment). Expansion Cohort: Day 1 and Day 8 at predose; 0.5 to 4 hr and 8 to 12 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose
Mean area under the concentration-time curve from zero time to time of last quantifiable concentration (AUC[0-t]) for E7046 and its metabolite ER-888188 in plasma | Day 1, Day 8, Week 3, Week 7
  Dose-Escalation: Day 1 and Day 8 at predose (0 hr); 0.5, 1, 2, 4, 6, 8, 10, and 24 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose (from participants on E7046 treatment). Expansion Cohort: Day 1 and Day 8 at predose; 0.5 to 4 hr and 8 to 12 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose
Mean area under the plasma concentration-time curve extrapolated to infinity (AUC0-inf) for E7046 and its metabolite ER-888188 in plasma | Day 1, Day 8, Week 3, Week 7
  Dose-Escalation: Day 1 and Day 8 at predose (0 hr); 0.5, 1, 2, 4, 6, 8, 10, and 24 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose (from participants on E7046 treatment). Expansion Cohort: Day 1 and Day 8 at predose; 0.5 to 4 hr and 8 to 12 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose
Mean terminal elimination half-life (t1/2) of E7046 and its metabolite ER-888188 in plasma | Day 1, Day 8, Week 3, Week 7
  Dose-Escalation: Day 1 and Day 8 at predose (0 hr); 0.5, 1, 2, 4, 6, 8, 10, and 24 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose (from participants on E7046 treatment). Expansion Cohort: Day 1 and Day 8 at predose; 0.5 to 4 hr and 8 to 12 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose
Mean accumulation ratio (Rac) of E7046 and its metabolite ER-888188 in plasma | Day 1, Day 8, Week 3, Week 7
  Dose-Escalation: Day 1 and Day 8 at predose (0 hr); 0.5, 1, 2, 4, 6, 8, 10, and 24 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose (from participants on E7046 treatment). Expansion Cohort: Day 1 and Day 8 at predose; 0.5 to 4 hr and 8 to 12 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose
Mean peak-trough fluctuation (PTF) of E7046 and its metabolite ER-888188 in plasma | Day 1, Day 8, Week 3, Week 7
  Dose-Escalation: Day 1 and Day 8 at predose (0 hr); 0.5, 1, 2, 4, 6, 8, 10, and 24 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose (from participants on E7046 treatment). Expansion Cohort: Day 1 and Day 8 at predose; 0.5 to 4 hr and 8 to 12 hr postdose. Week 3 and Week 7 at predose; 0.5 to 4 hr and 8 to 12 hr postdose

CONTACTS AND LOCATIONS:
Locations (5):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Weill Cornell, New York, New York
- Marie-Skodowska Curie Cancer Centre, Warsaw, Poland
- United Kingdom (2):
  - The Christie, Manchester
  - Mount Vernon Hospital, Northwood

IPD SHARING:
Plan to Share IPD: No